CLINICAL TRIAL: NCT05033730
Title: Comparative Study Between VolumeControlled Ventilation and FlowControlled Ventilation Through Ultra-thin Tube in Upper Airway Surgery
Brief Title: Comparison Between VCV and FCV Through Ultra-thin Tube in Upper Airway Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-20-164; MRC-01-20-164 (Other: Hamad Medical Corporation)
Record Dates: First submitted 2021-07-28; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-07

CONDITIONS: Ventilation Therapy; Complications; Trachea
Keywords: Flow Controlled Ventilation,; Tritube,; Volume Controlled Ventilation,
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care: Control (Group A) (No Intervention): Patients who are scheduled for elective surgical upper airway surgery will be given General Anesthesia by an anesthesiologist who is the principal investigator and the surgical procedures will be done by the same ENT surgeon. IV Induction of Anesthesia with Propofol Target controlled infusion (TCI), Remifentanil Target controlled infusion (TCI) and Rocuronium (0.5mg/Kg) for muscle relaxation. The airway will be secured with cuffed endotracheal tube after direct laryngoscopy. After intubation by a Suitable size Endotracheal tube, they will be mechanically ventilated using Volume Controlled Ventilation (VCV) with 40% Oxygen and minute ventilation adjusted to keep ETCO2 of 40 mmHg or less, and a PEEP of 5 cmH2O.
- Intervention Group: (Group B) (Experimental): General Anesthesia will be induced with IV Induction of Anesthesia by an anesthesiologist with Propofol (Target controlled infusion), Remifentanil (Target controlled infusion), and Rocuronium (0.5mg/Kg) for muscle relaxation. The airway will be secured with cuffed Tritube after direct laryngoscopy. They will be mechanically ventilated using Flow Controlled Ventilation (FCV) with 40% Oxygen, Flow rate:13L/Min., Peak Airway Pressure (15 cmH2O), and a PEEP of (5 cmH2O) to keep ETCO2 of 40 mmHg or less. The anesthesia will be maintained with Intravenous Infusion of Propofol, Remifentanil (TCI) to keep BIS 40-60.
  Interventions: Device: Flow Controlled Ventilation

INTERVENTIONS:
Device: Flow Controlled Ventilation — Mechanically ventilated using Flow Controlled Ventilation (FCV)
  Arms: Intervention Group: (Group B)

SUMMARY:
Ventilation through the small endotracheal tube is not an uncommon situation. The indications for it differ from elective upper airway surgery to emergency ventilation through needle cricothyrotomy. Conventionally, ventilation through small endotracheal tubes has been challenging by jet ventilation with subsequent risk of barotrauma and inadequate gas exchange. Expiration during jet ventilation occurs passively.

DETAILED DESCRIPTION:
Upper airway endoscopy (micro laryngoscopy (MLS), pan endoscopy) is a minor upper airway procedure needing short duration general anesthesia, small calibrate endotracheal tube and manipulation of the airway. Because of airway manipulation and the surgery involves the airway, which is being shared with the anesthesiologist, there is a risk of interruption of ventilation, oxygenation and loss of airway in addition to inherent complications of surgery.

Methods:

After the patients will receive information about the study and informed consent will be taken. The patients will be randomized. In the control group, (group A) ventilation will be performed according to the routine big endotracheal tube. In the treatment group (group B), the ultra-thin ventilation tube will be placed using laryngoscopy. All other treatment will be unchanged. Data collection will be started 5 min after the initiation of the study. Demographic data, Past medical history, and examinations data will be collected after acceptance of the patient to be enrolled into the study and other ventilation parameters will be collected 5 min after the start of the the study which is Skin incision Primary endpoint is; to evaluate whether the Flow Controlled Ventilation (FCV) can also achieve adequate oxygenation and ventilation through small tube or not.

ELIGIBILITY:
Inclusion Criteria:

* Adult population of both sex (ASA I, II).
* Between18-65 years of age.
* Patients for the upper airway.
* Patients need intubation/invasive mechanical ventilation.

Exclusion Criteria:

* ASA >II
* Advanced Respiratory disease.
* Advanced cardiovascular disease.
* Smokers.
* Pregnancy.
* Recent upper airway trauma.
* Age less than 18 years or more than 65 years.
* Patients BMI of more than 35
* Refuse to sign the consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of dynamic chest wall compliance (mL/mbar) | During study time intra-operatively
  Dynamic chest wall compliance changes due to Flow Controlled Ventilation (FCV) in comparison to routine Volume Controlled Ventilation(VCV)
Airway Resistance (mbar*s/L) | During procedure time and intra-operatively
  This measures the airway resistance changes due to Flow Controlled Ventilation (FCV) in comparison to the traditional Volume Controlled Ventilation(VCV)

SECONDARY OUTCOMES:
Oxygen concentration (SPaO2)and tension(PaO2) in the blood (% and mmHg respectively) | Intra-operatively during procedure time
  This will measure the patient oxygenation during intervention in both studied groups and using the arterial blood gases
Carbon dioxide in the blood (PaCO2) and the trachea (ECO2) mmHg. | During surgical procedure intra-operatively
  This measures the patient ventilation during intervention in both studied groups using capnogram and arterial blood gases
Postoperative sore throat according the Visual Analogue Scale (VAS) | After surgical procedure (2 and 24) hours.
  Postoperative sore throat after 2 and 24 hours using the VAS score (0-10). (Zero=no pain and 10 = for the most sever pain.
Kink of the small size tube (Tritube) (Yes/No) | During surgical procedure
  Kink of the small (Tritube) (using machine alarms for obstruction and visual inspection) so will be (yes) for partial or complete obstruction and (no) for the absence of obstruction)
Surgeon satisfaction instance scale (1-5) | During surgical procedure
  the Surgeon satisfaction score according the space free for the surgery which range from (1= poor, 2= medium, 3= good, 4= very good, and 5= excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Shallik, M.D., Principal Investigator — Hamad Medical Corporation - HMC
Locations (1):
- ACC&HGH, Hamad Medical Corporation, Doha, Doah, Qatar

IPD SHARING:
Plan to Share IPD: Yes
I will Share IPD data after IRB approval
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After IRB approval directly
Access Criteria: Website

REFERENCES:
- [Background] Schmidt J, Gunther F, Weber J, Wirth S, Brandes I, Barnes T, Zarbock A, Schumann S, Enk D. Flow-controlled ventilation during ear, nose and throat surgery: A prospective observational study. Eur J Anaesthesiol. 2019 May;36(5):327-334. doi: 10.1097/EJA.0000000000000967. PMID 30730422
- [Result] Putz L, Mayne A, Dincq AS. Jet Ventilation during Rigid Bronchoscopy in Adults: A Focused Review. Biomed Res Int. 2016;2016:4234861. doi: 10.1155/2016/4234861. Epub 2016 Oct 26. PMID 27847813
- [Result] Jeyarajah K, Ahmad I. Awake tracheal placement of the Tritube under flexible bronchoscopic guidance. Anaesthesia Cases. 2018 Jul;6(2):1-5.